CLINICAL TRIAL: NCT00518427
Title: A Multicenter Clinical Trial to Evaluate Quality of Life in Patients With Type 2 Diabetes Before and After Changing Therapy to a Combination of Insulin Glargine and Oral Antidiabetic Drugs in a Real Life Situation
Brief Title: Evaluate Quality of Life in Type 2 Diabetes, Before and After Change to Insuline Glargine
Acronym: QoL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4057; Eudract #: 2005-000959-15
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

ARMS (1):
- 1 (Experimental): insulin glargine
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — Lantus (insulin glargine [rDNA origin] injection), individual dosing , subcutaneous injection, 100 IU/ml.
  Duration of treatment will be judge by the investigator. Last QoL assessed in the study will be 9 months after start of glargine treatment.

SUMMARY:
Primary objective:

To assess quality of Life (QoL) changes and treatment satisfaction in a real life situation in patients with Type 2 diabetes inadequately controlled on a combination of oral antidiabetic drugs (OAD) plus Neutral Protamine Hagedrone (NHP) insulin treatment that are switched to insulin glargine.

Secondary objective:

To determine:

change in HbA1c, comparision of the incidence of symptomatic hypoglycemia and severe hypoglycemia before and after introduction of insulin glargine, change in weight, change in insulin dose.

ELIGIBILITY:
lists of inclusion and exclusion criteria:

Inclusion Criteria:

* Patients with type 2diabetes inadequately controlled on a combination of OAD + NPH insulin for more than three months
* Stable OAD therapy for at least three months, according to the following specified daily dose: glibenclamide> 3, 5 mg, glipizid >5 mg, glimeperid >2mg, metformin>1000 mg, acarbose >150 mg
* HbA1c > 7,0%
* Ability to perform QoL assessment
* Body Mass Indes: women <30 and men <32

Exlusion criteria:

* Autoimmune diabetes, as defined by WHO
* Ongoing treatment with tiasolidindion drug
* Retinopathy with surgical treatment during preceding three months of study entry or requiring treatment within three months after study entry
* Drug abuse
* Hypersensitivity to insulin glagine excipients

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The fear of hypoglycaemia scale (HFS) | before the switch to insulin glargine and at 3 and 9 months of follow up.
12 - Item Well-Being Questionnaaire (WBQ12) | before the switch to insulin glargine and at 3 and 9 months of follow up.
Glycaemic controll will be asessed by HbA1c values | week 12 and week 40

SECONDARY OUTCOMES:
Incidence of symptomatic hypoglycemia and severe hypoglycemia | sreening to follow-up phases

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Olsson-Birgersson, Study Director — sanofi-aventis, Sweden
Locations (1):
- Sanofi-Aventis Administrative Office, Bromma, Sweden